CLINICAL TRIAL: NCT01766050
Title: An Open-label, Single-sequence Study of the Effect of Belatacept on the Pharmacokinetics of Caffeine, Losartan, Omeprazole, Dextromethorphan, and Midazolam Administered as "Inje Cocktail" in Healthy Subjects
Brief Title: Study to Evaluate Effect of Belatacept on Pharmacokinetics of Inje Cocktail in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IM103-151
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Transplant Rejection
MeSH Terms: interventions — Caffeine; Losartan; Omeprazole; Dextromethorphan; Midazolam; Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm: Inje Cocktail + Belatacept (Experimental): Inje Cocktail consisting of (200 mg Caffeine, 50 mg losartan tablet, 40 mg Omeprazole capsule, 30 mg Dextromethorphan capsule and 5 mg Midazolam oral syrup) administered on Days 1, 4, 7 and 11
  Belatacept 10 mg/kg Intravenous (IV) solution, administered on Day 4
  Interventions: Drug: Caffeine; Drug: Losartan; Drug: Omeprazole; Drug: Dextromethorphan; Drug: Midazolam; Biological: Belatacept

INTERVENTIONS:
Drug: Caffeine
Drug: Losartan
Drug: Omeprazole
Drug: Dextromethorphan
Drug: Midazolam
Biological: Belatacept
  Other Names: Nulojix; BMS-224818

SUMMARY:
The purpose of this study is to determine the effects of belatacept on the pharmacokinetics of caffeine, losartan, omeprazole, dextromethorphan and midazolam

ELIGIBILITY:
Inclusion Criteria:

* BMI 18 to 30 kg/m2
* Men and women ages 18 to 45

Exclusion Criteria:

* Active tuberculosis
* Any recent infection requiring antibiotic treatment within 4 weeks of dosing
* Positive urine screen for drugs of abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Healthcare Discoveries, Llc D/B/A Icon Development Solutions, San Antonio, Texas, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated January 2013 and completed April 2013. Participants (healthy volunteers) checked into a clinical pharmacology unit (CPU) on Day -1 for screening.
Pre-assignment Details: 45 were enrolled and 22 dosed with study drug. Reasons for not dosing: 5 withdrew consent, 1 lost to follow up, 1 poor/non-compliance, 15 no longer met study criteria, and 1 other.
Groups:
- Inje Cocktail Alone and Inje Cocktail Plus Belatacept: Single oral doses of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) were administered on Days 1, 4, 7 and 11. A single 10 mg/kg intravenous (IV) infusion of belatacept over 30 minutes was administered on Day 4.
Period: Overall Study
Arm/Group | Inje Cocktail Alone and Inje Cocktail Plus Belatacept
Started | 22
Completed | 18
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All participants who received study drug.
Arm/Group | Inje Cocktail Alone and Inje Cocktail Plus Belatacept
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (5.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — body mass index (BMI): weight in kilograms (kg)/[height in meters (m)]2
  kg/m^2 | 24.62 (2.886)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric Mean Maximum Drug Concentration (Cmax) of Midazolam With and Without the Coadministration of Belatacept - Pharmacokinetic (PK) Evaluable Population
Description: Samples for the assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) and their metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Adjusted geometric mean for midazolam with and without belatacept, along with adjusted geometric mean ratios for Days 4, 7, and 11 versus Day 1, respectively, are presented. Cmax measured in nanograms per milliliter (ng/mL). Inje cocktail components (Midazolam) measured using High Performance Liquid Chromatography (HPLC) with Tandem Mass Spectrometry (MS/MS) Detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: Participants who received any study drug and had at least 1 adequate Pharmacokinetic (PK) profile for any Inje cocktail analytes (parent or metabolite).
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Day 1 Inje Cocktail: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Day 1.
- Day 4 Inje Cocktail Plus Belatacept: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Day 4. A single 10 mg/kg intravenous (IV) infusion of belatacept over 30 minutes was administered only on Day 4.
- Day 7 Inje Cocktail: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Day 7.
- Day 11 Inje Cocktail: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Day 11.
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ng/mL | 24.376 (42) [21.117 to 28.137] | 24.152 [20.632 to 28.271] | 22.211 [19.131 to 25.787] | 24.220 [20.835 to 28.154]
Statistical Analysis 1: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.991, 90% CI 2-sided [0.898 to 1.093]
Statistical Analysis 2: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.911, 90% CI 2-sided [0.830 to 1.000]
Statistical Analysis 3: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.994, 90% CI 2-sided [0.885 to 1.116]

2. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of the Inje Cocktail Components (Midazolam, Losartan, Omeprazole, Dextromethorphan, and Caffeine) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. The poor metabolizer of CYP2D6 was excluded from summary of dextromethorphan parameters. Inje cocktail components were each measured using HPLC with MS/MS detection. Tmax was measured in hours (h).
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Measure: Median (Full Range); unit: h
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
h
  Midazolam (N=22,21,21,20) | 0.50 [0.50 to 1.50] | 0.50 [0.50 to 1.50] | 0.50 [0.50 to 1.50] | 1.0 [0.50 to 1.03]
  Losartan (N= 22, 21, 21, 20) | 1.52 [0.50 to 3.00] | 2.00 [0.50 to 4.00] | 1.50 [0.50 to 3.00] | 1.50 [0.50 to 3.00]
  Omeprazole (N=22,21,21,20) | 2.00 [1.50 to 4.00] | 3.00 [1.00 to 8.05] | 3.00 [1.00 to 5.00] | 3.00 [1.00 to 12.00]
  Dextromethorphan (N=21, 19, 19, 19) | 3.00 [1.00 to 6.00] | 3.00 [1.50 to 6.00] | 3.00 [1.50 to 5.15] | 3.00 [1.00 to 6.00]
  Caffeine (N= 22,21,21,18) | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 3.00] | 1.50 [0.50 to 4.00] | 1.50 [0.50 to 2.00]

3. Secondary Outcome: Plasma Half-Life (T-HALF) of the Inje Cocktail Components (Midazolam, Losartan, Omeprazole, Dextromethorphan, and Caffeine) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. The poor metabolizer of CYP2D6 was excluded from summary of dextromethorphan parameters. Inje cocktail components were each measured using HPLC with MS/MS detection. T-HALF was measured in hours (h).
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: Evaluable PK population: Participants who received any study drug and had at least 1 adequate PK profile for any Inje cocktail analytes (parent or metabolite).
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
h
  Midazolam (N=22, 21, 21, 20) | 4.01 (1.86) | 4.43 (1.89) | 4.27 (1.88) | 4.05 (1.61)
  Losartan (N=22, 21, 21, 20) | 2.96 (1.29) | 2.56 (1.31) | 3.30 (1.49) | 2.87 (1.52)
  Omeprazole (N= 22, 19, 21, 18) | 1.19 (0.497) | 1.39 (0.569) | 1.28 (0.470) | 1.36 (0.907)
  Dextromethorphan (N=18, 17, 18, 15) | 6.76 (2.09) | 6.98 (2.67) | 6.33 (1.69) | 6.70 (2.29)
  Caffeine (N=22, 21, 21, 18) | 5.61 (1.87) | 5.71 (2.01) | 6.17 (2.29) | 6.03 (2.13)

4. Secondary Outcome: Apparent Total Body Clearance (CLT/F) of the Inje Cocktail Components (Midazolam, Losartan, Omeprazole, Dextromethorphan and Caffeine) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. The poor metabolizer of CYP2D6 was excluded from summary of dextromethorphan parameters. Inje cocktail components were each measured using HPLC with MS/MS detection. CLT/F was measured as liters/hour (L/h)
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
L/h
  Midazolam (N=22, 21, 21, 20) | 73.8 (49) | 71.3 (48) | 77.3 (50) | 71.4 (51)
  Losartan (N=22, 21, 21, 20) | 148 (37) | 146 (36) | 146 (34) | 151 (44)
  Omeprazole (N=22, 19, 21, 18) | 29.2 (66) | 23.7 (72) | 24.7 (79) | 25.3 (69)
  Dextromethorphan (N=18,17,18,18) | 3916 (85) | 4247 (84) | 4264 (126) | 3968 (107)
  Caffeine (N=22, 21, 21, 18) | 4.99 (34) | 5.30 (32) | 4.97 (36) | 4.83 (36)

5. Secondary Outcome: Cmax of Inje Cocktail Metabolites (1'-Hydroxy-Midazolam, E-3174, 5-Hydroxyomeprazole, Dextrorphan, and Paraxanthine) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Samples for assessment of plasma concentrations of Inje cocktail component metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. The poor metabolizer of CYP2D6 was excluded from summary of Dextrorphan parameters. Inje cocktail component metabolites were each measured using HPLC with MS/MS detection. Cmax was measured in ng/mL.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Day 4 Inje Cocktail Plus Belatacept: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Days 4. A single 10 mg/kg intravenous (IV) infusion of belatacept over 30 minutes was administered only on Day 4.
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ng/mL
  1'-Hydroxy-Midazolam (N=22, 21, 21, 20) | 11.1 (40) | 11.9 (40) | 11.4 (38) | 12.3 (36)
  E-3174 (N=22, 21, 21, 20) | 262 (37) | 276 (33) | 300 (33) | 291 (41)
  5-Hydroxyomeprazole (N=22, 21, 21, 20) | 335 (41) | 360 (40) | 332 (38) | 337 (38)
  Dextrorphan (N=21,20,20,19) | 342 (30) | 324 (32) | 312 (31) | 331 (35)
  Paraxanthine (N=17,19,18,18) | 1291 (15) | 1367 (12) | 1320 (13) | 1358 (15)

6. Secondary Outcome: AUC(0-T) of Inje Cocktail Component Metabolites (1'-Hydroxy-Midazolam, E-3174, 5-Hydroxyomeprazole, Dextrorphan, and Paraxanthine) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Area under the plasma concentration-time curve from zero to the last time of the last quantifiable concentration [AUC(0-T)] was measured in ng*h/mL. Samples for assessment of plasma concentrations of Inje cocktail components metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. The poor metabolizer of CYP2D6 was excluded from summary of Dextrorphan parameters. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ng*h/mL
  1'-hydroxy-midazolam (N=22, 21, 21, 20) | 28.9 (39) | 31.8 (30) | 32.5 (32) | 33.6 (27)
  E-3174 (N= 22,21,21,20) | 1995 (32) | 1999 (29) | 2089 (30) | 2072 (37)
  5-hydroxyomeprazole (N=22,21,21,20) | 997 (36) | 967 (33) | 929 (35) | 995 (35)
  dextrorphan (N=21,20,20,19) | 1636 (27) | 1570 (26) | 1519 (27) | 1644 (26)
  paraxanthine (N=17,19,18,18) | 20592 (15) | 21077 (16) | 20680 (18) | 21353 (20)

7. Secondary Outcome: AUC(INF) of Inje Cocktail Component Metabolites (1'-Hydroxy-Midazolam, E-3174, 5-Hydroxyomeprazole, Dextrorphan, and Paraxanthine) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] was measured in ng*h/mL. Samples for assessment of plasma concentrations of Inje cocktail components metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. The poor metabolizer of CYP2D6 was excluded from summary of Dextrorphan parameters. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ng*h/mL
  1'-hydroxy-midazolam (N=22,21,20,20) | 30.5 (38) | 33.8 (32) | 32.9 (27) | 35.1 (27)
  E-3174 (N=22,20,21,20) | 2103 (32) | 2060 (29) | 2187 (31) | 2182 (38)
  5-hydroxyomeprazole (N=22,20,21,17 | 1010 (36) | 990 (34) | 938 (35) | 1063 (32)
  dextrorphan (N=21,20,20,19) | 1679 (25) | 1610 (25) | 1562 (26) | 1682 (25)
  paraxanthine (N=7,8,6,6) | 22401 (18) | 22905 (24) | 22063 (12) | 21874 (20)

8. Secondary Outcome: Tmax of Inje Cocktail Component Metabolites (1'-Hydroxy-Midazolam, E-3174, 5-Hydroxyomeprazole, Dextrorphan, and Paraxanthine) With and Without the Coadministration of Belatacept - PK Evaluable Population
Description: Samples for assessment of plasma concentrations of Inje cocktail components metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. The poor metabolizer of CYP2D6 was excluded from summary of Dextrorphan parameters. Inje cocktail components were each measured using HPLC with MS/MS detection. Time of maximum observed plasma concentration (Tmax) was measured in hours (h).
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Median (Full Range); unit: h
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
h
  1'-Hydroxy-Midazolam (N=22,21,21,20) | 1.00 [0.50 to 1.50] | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 1.50] | 1.00 [0.50 to 1.50]
  E-3174 (N=22, 21, 21, 20) | 4.00 [3.00 to 5.03] | 4.00 [2.00 to 8.00] | 4.00 [3.00 to 5.15] | 4.00 [3.00 to 6.02]
  5-Hydroxyomeprazole (N=22,21,21,20) | 2.00 [1.50 to 5.00] | 3.00 [1.00 to 8.05] | 3.00 [1.00 to 5.00] | 2.53 [1.00 to 12.00]
  Dextrorphan (N=21,20,20,19) | 2.00 [1.50 to 4.00] | 2.00 [1.50 to 4.00] | 2.00 [1.50 to 3.00] | 2.00 [1.50 to 4.00]
  Paraxanthine (N=17, 19, 18, 18) | 8.00 [3.00 to 12.02] | 8.00 [5.00 to 12.00] | 8.00 [4.0 to 12.00] | 8.00 [4.00 to 12.00]

9. Secondary Outcome: T-HALF of Inje Cocktail Component Metabolites (1'-Hydroxy-Midazolam, E-3174, 5-Hydroxyomeprazole, Dextrorphan, and Paraxanthine) With and Without the Coadministration of Belatacept - PK Evaluable Population
Description: Plasma half-life (T-HALF) was measured in hours (h). Samples for assessment of plasma concentrations of Inje cocktail components metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. The poor metabolizer of CYP2D6 was excluded from summary of Dextrorphan parameters. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
h
  1'-Hydroxy-Midazolam (N=22,21,20,20) | 5.29 (2.98) | 6.35 (3.60) | 5.61 (3.47) | 5.31 (2.65)
  E-3174 (N=22, 20, 21, 20) | 4.86 (0.749) | 4.57 (0.757) | 4.75 (0.757) | 4.88 (0.690)
  5-Hydroxyomeprazole (N=22,20,21,17) | 1.43 (0.308) | 1.55 (0.397) | 1.52 (0.371) | 1.54 (0.624)
  Dextrorphan (N=21,20,20,19) | 4.26 (1.60) | 4.36 (1.46) | 4.23 (1.13) | 4.08 (0.999)
  Paraxanthine (N=7,8,6,6) | 7.33 (1.91) | 6.86 (1.71) | 7.33 (1.55) | 7.44 (2.67)

10. Secondary Outcome: Ratio of Paraxanthine AUC(0-T) to Caffeine AUC(0-T) and Paraxanthine AUC (INF) to Caffeine AUC (INF), Corrected for Molecular Weight [MR_AUC(0-T) and MR_AUC (INF)] With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Metabolite (paraxanthine) to parent (caffeine) ratio was corrected for molecular weight. AUC (0-T) and AUC (INF) measured in ng*h/mL. Samples for assessment of plasma concentrations of Inje cocktail components and the metabolites of those components were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 17 | 19 | 18 | 18
ratio
  MR_AUC(0-T) ratio; N=17,19,18,18 | 0.627 (24) | 0.677 (17) | 0.635 (20) | 0.603 (21)
  MR_AUC(INF) ratio; N=7, 8, 6, 6 | 0.827 (15) | 0.827 (8) | 0.799 (14) | 0.781 (12)

11. Secondary Outcome: Ratio of Paraxanthine (Cmax) to Caffeine (Cmax), Corrected for Molecular Weight (MR_Cmax) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Metabolite (paraxanthine) to parent (caffeine) ratio was corrected for molecular weight. Cmax measured in ng/mL. Samples for assessment of plasma concentrations of Inje cocktail components and their metabolites were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Groups:
- Day 4 Inje Cocktail Plus Belatacept: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Day 4. A single 10 mg/kg IV infusion of belatacept over 30 minutes was administered only on Day 4.
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 17 | 19 | 18 | 18
ratio | 0.303 (22) | 0.337 (15) | 0.333 (23) | 0.323 (20)

12. Secondary Outcome: Ratio of E-3174 AUC(0-T) to Losartan AUC(0-T) and E3174 AUC (INF) to Losartan AUC (INF) Corrected for Molecular Weight [MR_AUC(0-T), MR_AUC(INF)] With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Metabolite (E-3174) to parent (losartan) ratio was corrected for molecular weight. AUC (0-T) and AUC (INF) measured in ng*h/mL. Samples for assessment of plasma concentrations of Inje cocktail components and the metabolites of those components were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ratio
  MR_AUC (0-T) ratio; N=22,21,21,20 | 5.81 (32) | 5.75 (33) | 5.99 (33) | 6.17 (33)
  MR_AUC (INF) ratio; N=22,20,21,20 | 6.02 (30) | 5.99 (32) | 6.16 (32) | 6.37 (31)

13. Secondary Outcome: Ratio of E-3174 (Cmax) to Losartan (Cmax), Corrected for Molecular Weight (MR_Cmax) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Metabolite (E-3174) to parent (losartan) ratio was corrected for molecular weight. Cmax measured in ng/mL. Samples for assessment of plasma concentrations of Inje cocktail components and the metabolites of those components were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ratio | 2.31 (39) | 2.24 (45) | 2.26 (43) | 2.26 (45)

14. Secondary Outcome: Ratio of 5-Hydroxyomeprazole AUC(0-T) to Omeprazole AUC(0-T) and 5-Hydroxyomeprazole AUC(INF) to Omeprazole AUC(INF) , Corrected for Molecular Weight [MR_AUC(0-T), MR_AUC(INF)] With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Metabolite (5-Hydroxyomeprazole) to parent (omeprazole) ratio was corrected for molecular weight. AUC (0-T) and AUC (INF) measured in ng*h/mL. Samples for assessment of plasma concentrations of Inje cocktail components and the metabolites of those components were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ratio
  MR_AUC (0-T) ratio; N=22,21,21,20 | 0.700 (57) | 0.609 (66) | 0.551 (70) | 0.610 (66)
  MR_AUC (INF) ratio; N=22,19,21,17 | 0.705 (56) | 0.558 (61) | 0.553 (69) | 0.679 (62)

15. Secondary Outcome: Ratio of 5-Hydroxyomeprazole (Cmax) to Omeprazole (Cmax), Corrected for Molecular Weight (MR_Cmax) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Metabolite (5-hydroxyomeprazole) to parent (omeprazole) ratio was corrected for molecular weight. Cmax measured in ng/mL. Samples for assessment of plasma concentrations of Inje cocktail components and the metabolites of those components were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ratio | 0.548 (54) | 0.471 (60) | 0.424 (65) | 0.478 (59)

16. Secondary Outcome: Ratio of 5-Dextrorphan AUC(0-T) to Dextromethorphan AUC(0-T) and 5-Dextrorphan AUC(INF) to Dextromethorphan AUC(INF), Corrected for Molecular Weight [MR_AUC(0-T), MR_AUC (INF)] With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Metabolite (5-dextrorphan ) to parent (dextromethorphan) ratio was corrected for molecular weight. AUC (0-T) and AUC (INF) measured in ng*h/mL. Samples for assessment of plasma concentrations of Inje cocktail components and the metabolites of those components were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. The poor metabolizer of CYP2D6 was excluded from summary of Dextrorphan parameters. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 21 | 20 | 20 | 19
ratio
  MR_AUC (0-T) ratio; N=21,20,20,19 | 201 (103) | 200 (94) | 177 (124) | 193 (99)
  MR_AUC (INF) ratio; N=18,17,18,15 | 173 (95) | 177 (90) | 170 (122) | 173 (102)

17. Secondary Outcome: Ratio of 5-Dextrorphan (Cmax) to Dextromethorphan (Cmax), Corrected for Molecular Weight (MR_Cmax) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Metabolite (5-dextrorphan) to parent (dextromethorphan) ratio was corrected for molecular weight. Cmax measured in ng/mL. Samples for assessment of plasma concentrations of Inje cocktail components and the metabolites of those components were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. The poor metabolizer of CYP2D6 was excluded from summary of Dextrorphan parameters. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 21 | 20 | 20 | 19
ratio | 280 (107) | 303 (99) | 275 (88) | 303 (84)

18. Secondary Outcome: Ratio of 1'-Hydroxy-Midazolam AUC(0-T) to Midazolam AUC(0-T) and 1'-Hydroxy-Midazolam AUC(INF) to Midazolam AUC(INF), Corrected for Molecular Weight [MR_AUC(0-T), MR_AUC (INF)] With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Metabolite (1'-hydroxy-midazolam) to parent (midazolam) ratio was corrected for molecular weight. AUC (0-T) and AUC (INF) measured in ng*h/mL. Samples for assessment of plasma concentrations of Inje cocktail components and the metabolites of those components were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ratio
  MR_AUC (0-T) ratio; N=22, 21, 21, 20 | 0.421 (56) | 0.447 (46) | 0.495 (55) | 0.472 (55)
  MR_(INF) ratio; N=22, 21, 20, 20 | 0.428 (57) | 0.460 (47) | 0.479 (52) | 0.478 (55)

19. Primary Outcome: Adjusted Geometric Mean Area Under the Concentration Time Curve (AUC) From Zero to Last Concentration (0-T) and AUC Extrapolated to Infinity (INF) of Midazolam With and Without the Coadministration of Belatacept - Pharmacokinetic (PK) Evaluable Population
Description: AUC(0-T): area under the plasma concentration-time curve from zero to the last time of the last quantifiable concentration and AUC (INF): AUC from time zero extrapolated to infinite time were measured in ng*h/mL. Samples for the assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) and their metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Adjusted geometric mean for midazolam with and without belatacept, along with adjusted geometric mean ratios for Days 4, 7, and 11 versus Day 1, respectively, are presented. Midazolam measured using HPLC with MS/MS Detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7and 11
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ng*h/mL
  AUC (0-T);N=22, 21, 21, 20) | 65.548 [53.271 to 80.655] | 68.833 [57.008 to 83.111] | 63.303 [52.240 to 76.707] | 67.717 [56.128 to 81.697]
  AUC (INF);N=22, 21, 21, 20) | 67.743 [54.839 to 83.683] | 71.039 [58.555 to 86.186] | 65.555 [54.019 to 79.554] | 69.841 [57.771 to 84.433]
Statistical Analysis 1: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.050, 90% CI 2-sided [0.976 to 1.130]
Statistical Analysis 2: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 0.966, 90% CI 2-sided [0.889 to 1.049]
Statistical Analysis 3: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.033, 90% CI 2-sided [0.950 to 1.123]
Statistical Analysis 4: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.049, 90% CI 2-sided [0.975 to 1.127]
Statistical Analysis 5: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 0.968, 90% CI 2-sided [0.892 to 1.049]
Statistical Analysis 6: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; AUC(INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.031, 90% CI 2-sided [0.948 to 1.121]

20. Primary Outcome: Adjusted Geometric Mean Cmax of Losartan With and Without the Coadministration of Belatacept - PK Evaluable Population
Description: Cmax measured in ng/mL. Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) and their metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Adjusted geometric mean for losartan with and without belatacept, along with adjusted geometric mean ratios for Days 4, 7, and 11 versus Day 1, respectively, are presented. Inje cocktail components (losartan) measured using HPLC with MS/MS Detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Day 4 Inje Cocktail Plus Belatacept: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Day 4. A single 10 mg/kg intravenous (IV) infusion of belatacept over 30 minutes was administered on Day 4.
- Day 11 Inje Cocktail: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Day 1, 4, 7 and 11.
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ng/mL | 119.789 [89.629 to 134.485] | 118.663 [97.209 to 144.850] | 127.184 [105.467 to 153.373] | 126.461 [101.676 to 157.288]
Statistical Analysis 1: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.991, 90% CI 2-sided [0.898 to 1.093]
Statistical Analysis 2: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.911, 90% CI 2-sided [0.830 to 1.000]
Statistical Analysis 3: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.994, 90% CI 2-sided [0.885 to 1.116]

21. Primary Outcome: Adjusted Geometric Mean AUC (0-T) and AUC (INF) of Losartan With and Without the Coadministration of Belatacept - Pharmacokinetic (PK) Evaluable Population
Description: AUC (0-T): area under the concentration curve from time 0 to the time of the last quantifiable concentration and AUC (INF) extrapolated to infinity were measured in ng*h/mL. Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) and their metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Adjusted geometric mean for losartan with and without belatacept, along with adjusted geometric mean ratios for Days 4, 7, and 11 versus Day 1, respectively, are presented. Inje cocktail components (losartan) measured using HPLC with MS/MS Detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ng*h/mL
  AUC (0-T) N=22, 21, 21, 20) | 332.191 [283.753 to 388.898] | 336.531 [291.278 to 388.815] | 337.487 [295.482 to 385.462] | 332.400 [280.799 to 393.484]
  AUC (INF) N=22, 21, 21, 20) | 338.033 [289.143 to 395.189] | 341.644 [296.237 to 394.012] | 343.508 [301.494 to 391.378] | 338.646 [286.824 to 399.831]
Statistical Analysis 1: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.013, 90% CI 2-sided [0.944 to 1.088]
Statistical Analysis 2: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.016, 90% CI 2-sided [0.936 to 1.103]
Statistical Analysis 3: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.001, 90% CI 2-sided [0.893 to 1.121]
Statistical Analysis 4: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.011, 90% CI 2-sided [0.942 to 1.085]
Statistical Analysis 5: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.016, 90% CI 2-sided [0.938 to 1.101]
Statistical Analysis 6: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.002, 90% CI 2-sided [0.896 to 1.121]

22. Primary Outcome: Adjusted Geometric Mean Cmax of Omeprazole With and Without the Coadministration of Belatacept - Pharmacokinetic (PK) Evaluable Population
Description: Cmax: Maximum observed plasma concentration was measured in ng/mL. Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) and their metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Adjusted geometric mean for omeprazole with and without belatacept, along with adjusted geometric mean ratios for Days 4, 7, and 11 versus Day 1, respectively, are presented. Inje cocktail components (omeprazole) measured using HPLC with MS/MS Detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ng/mL | 583.047 [473.091 to 718.560] | 734.776 [587.280 to 919.316] | 753.126 [597.946 to 948.579] | 686.929 [555.590 to 849.315]
Statistical Analysis 1: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.260, 90% CI 2-sided [1.118 to 1.421]
Statistical Analysis 2: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.292, 90% CI 2-sided [1.090 to 1.531]
Statistical Analysis 3: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.178, 90% CI 2-sided [0.971 to 1.429]

23. Primary Outcome: Adjusted Geometric Mean AUC (0-T) and AUC (INF) of Omeprazole With and Without the Coadministration of Belatacept - Pharmacokinetic (PK) Evaluable Population
Description: AUC(0-T): Area under the plasma concentration-time curve from time zero zero to the time of the last quantifiable concentration and AUC (INF): AUC extrapolated to infinity were measured in ng*h/mL. Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) and their metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Adjusted geometric mean for omeprazole with and without belatacept, along with adjusted geometric mean ratios for Days 4, 7, and 11 versus Day 1, respectively, are presented. Inje cocktail components (omeprazole) measured using HPLC with MS/MS Detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Groups:
- Day 1 Inje Cocktail: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Days 1.
- Day 11 Inje Cocktail: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Day11.
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ng*h/mL
  AUC (0-T); (N= 22, 21, 21, 20) | 1361.024 [1066.457 to 1736.953] | 1577.017 [1200.238 to 2072.075] | 1671.173 [1278.936 to 2183.704] | 1653.491 [1264.315 to 2162.463]
  AUC (INF); (N= 22, 19, 21, 18) | 1368.593 [1072.836 to 1745.885] | 1632.455 [1251.956 to 2128.597] | 1679.693 [1286.299 to 2193.400] | 1779.717 [1380.250 to 2294.798]
Statistical Analysis 1: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.159, 90% CI 2-sided [1.056 to 1.272]
Statistical Analysis 2: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.228, 90% CI 2-sided [1.092 to 1.381]
Statistical Analysis 3: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.215, 90% CI 2-sided [1.047 to 1.410]
Statistical Analysis 4: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.193, 90% CI 2-sided [1.091 to 1.304]
Statistical Analysis 5: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.227, 90% CI 2-sided [1.093 to 1.379]
Statistical Analysis 6: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.300, 90% CI 2-sided [1.141 to 1.482]

24. Primary Outcome: Adjusted Geometric Mean Cmax of Dextromethorphan With and Without the Coadministration of Belatacept - PK Evaluable Population
Description: Cmax was measured in ng/mL. Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) and their metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Adjusted geometric mean for dextromethorphan with and without belatacept, along with adjusted geometric mean ratios for Days 4, 7, and 11 versus Day 1, respectively, are presented. The poor metabolizer of CYP2D6 was excluded from the statistical analysis. Inje cocktail components (dextromethorphan) measured using HPLC with MS/MS Detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 21 | 19 | 19 | 19
ng/mL | 0.927 [0.566 to 1.518] | 0.800 [0.512 to 1.250] | 0.855 [0.553 to 1.320] | 0.794 [0.490 to 1.286]
Statistical Analysis 1: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.863, 90% CI 2-sided [0.746 to 0.997]
Statistical Analysis 2: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.922, 90% CI 2-sided [0.793 to 1.071]
Statistical Analysis 3: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.856, 90% CI 2-sided [0.709 to 1.034]

25. Primary Outcome: Adjusted Geometric Mean AUC (0-T) and AUC (INF) of Dextromethorphan With and Without the Coadministration of Belatacept - PK Evaluable Population
Description: AUC(0-T): area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration and AUC (INF): AUC extrapolated to infinity, were measured as ng*h/mL. Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) and their metabolites (1'-hydroxy-midazolam, E-3174, 5-hydroxyomeprazole, dextrorphan, and paraxanthine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Adjusted geometric mean for dextromethorphan with and without belatacept, along with adjusted geometric mean ratios for Days 4, 7, and 11 versus Day 1, respectively, are presented. The poor metabolizer of CYP2D6 was excluded from the statistical analysis. Inje cocktail components (dextromethorphan) measured using HPLC with MS/MS Detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Groups:
- Day 1 Inje Cocktail: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Day1.
- Day 4 Inje Cocktail Plus Belatacept: Single oral dose of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) was administered on Day 4. A single 10 mg/kg IV infusion of belatacept over 30 minutes was administered on Day 4.
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 21 | 19 | 19 | 19
ng*h/mL
  AUC (0-T); N= 21, 19, 19, 19 | 6.176 [3.466 to 11.005] | 5.651 [3.305 to 9.661] | 6.195 [3.705 to 10.358] | 5.949 [3.465 to 10.215]
  AUC (INF); N= 18, 17, 18, 15 | 6.220 [3.743 to 10.337] | 5.455 [3.372 to 8.825] | 6.412 [4.200 to 9.790] | 6.359 [1.143 to 9.760]
Statistical Analysis 1: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 0.915, 90% CI 2-sided [0.817 to 1.024]
Statistical Analysis 2: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.003, 90% CI 2-sided [0.856 to 1.175]
Statistical Analysis 3: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 0.963, 90% CI 2-sided [0.821 to 1.130]
Statistical Analysis 4: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 0.877, 90% CI 2-sided [0.783 to 0.982]
Statistical Analysis 5: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.031, 90% CI 2-sided [0.885 to 1.200]
Statistical Analysis 6: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.022, 90% CI 2-sided [0.839 to 1.245]

26. Primary Outcome: Adjusted Geometric Mean Cmax of Caffeine With and Without the Coadministration of Belatacept - PK Evaluable Population
Description: Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Inje cocktail components were each measured using HPLC with MS/MS detection. Cmax was measured in ng/mL.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 18
ng/mL | 4696.505 [4252.803 to 5186.499] | 4450.019 [4172.484 to 4746.014] | 4332.326 [3993.257 to 4700.186] | 4479.687 [4141.210 to 4845.830]
Statistical Analysis 1: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.948, 90% CI 2-sided [0.880 to 1.021]
Statistical Analysis 2: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.922, 90% CI 2-sided [0.857 to 0.993]
Statistical Analysis 3: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.954, 90% CI 2-sided [0.885 to 1.028]

27. Primary Outcome: Adjusted Geometric Mean AUC (0-T) and AUC (INF) of Caffeine With and Without the Coadministration of Belatacept - PK Evaluable Population
Description: Samples for assessment of plasma concentrations of Inje cocktail components (midazolam, losartan, omeprazole, dextromethorphan and caffeine) were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Inje cocktail components were each measured using HPLC with MS/MS detection. AUC (0-T) and AUC (INF) were measured as ng*h/mL.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 18
ng*h/mL
  AUC (0-T); N= 22, 21, 21, 18 | 37394.5 [33103.4 to 42241.8] | 35200.3 [31255.9 to 39642.5] | 36853.4 [32319.8 to 42022.9] | 38407.0 [34164.2 to 43176.7]
  AUC (INF); N= 22, 21, 21, 18 | 40084.1 [34881.6 to 46062.5] | 37647.8 [32705.5 to 43336.9] | 40149.9 [34434.3 to 46814.1] | 41537.6 [36092.9 to 47803.7]
Statistical Analysis 1: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 0.941, 90% CI 2-sided [0.874 to 1.013]
Statistical Analysis 2: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 0.986, 90% CI 2-sided [0.902 to 1.076]
Statistical Analysis 3: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; AUC (0-T); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.027, 90% CI 2-sided [0.942 to 1.120]
Statistical Analysis 4: Comparison: Day 1 Inje Cocktail vs Day 4 Inje Cocktail Plus Belatacept; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 0.939, 90% CI 2-sided [0.868 to 1.017]
Statistical Analysis 5: Comparison: Day 1 Inje Cocktail vs Day 7 Inje Cocktail; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.002, 90% CI 2-sided [0.914 to 1.098]
Statistical Analysis 6: Comparison: Day 1 Inje Cocktail vs Day 11 Inje Cocktail; AUC (INF); Test type: Superiority or Other; Adjusted geometric mean ratio = 1.036, 90% CI 2-sided [0.940 to 1.142]

28. Secondary Outcome: Ratio of 1'-Hydroxy-Midazolam (Cmax) to Midazolam (Cmax), Corrected for Molecular Weight (MR_Cmax) With and Without Coadministration of Belatacept - PK Evaluable Population
Description: Metabolite (1'-hydroxy-midazolam) to parent (midazolam) ratio was corrected for molecular weight. Cmax measured in ng/mL. Samples for assessment of plasma concentrations of Inje cocktail components and the metabolites of those components were collected at time = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours relative to the dosing of belatacept on Day 4 and Inje cocktail dosing on Days 1, 4, 7, and 11, respectively. Inje cocktail components were each measured using HPLC with MS/MS detection.
Time Frame: Pre-dose to 24 hours after dose of the Inje Cocktail on Days 1, 4, 7 and 11
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
ratio | 0.432 (45) | 0.476 (44) | 0.497 (46) | 0.490 (46)

29. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Deaths, and AEs Leading to Discontinuation - All Treated Participants
Description: Adverse events were coded according to the Medical Dictionary for Regulatory Activities (MedDRA), version 15.1. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Events captured from Day 1 (pre-dose) to last day prior to discharge (Day 46 ±2). In the total group, a participant with an AE is only counted once (ie, data reflected in Days 1, 4, 7, and 11 below could be the same participant with an AE on multiple days of the study).
Time Frame: Day 1 to Day of discharge (Day 46±2)
Population: All participants who received any study medication.
Measure: Number; unit: participants
Groups:
- All Participants: Single oral doses of Inje Cocktail consisting of: caffeine (200 mg), losartan (50 mg tablet), omeprazole (40 mg delayed-release capsule), dextromethorphan (30 mg), and midazolam (5 mg oral syrup) were administered on Days 1, 4, 7 and 11. A single 10 mg/kg intravenous (IV) infusion of belatacept over 30 minutes was administered on Day 4.
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail | All Participants
Number analyzed (Participants) | 22 | 21 | 21 | 20 | 22
participants
  Adverse Events | 4 | 2 | 1 | 1 | 5
  SAEs | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0
  AEs leading to discontinuation | 0 | 0 | 1 | 0 | 1

30. Secondary Outcome: Number of Participants With Marked Serum Chemistry Laboratory Abnormalities - All Treated Participants
Description: Samples for laboratory tests were obtained at Screening visit, Day -1 or prior to dosing on Day 1, Days 3, 6, 10, 46, and at early termination, after 10 hours fasting. Upper limits of normal (ULN); Lower limits of normal (LLN); Pre-therapy (Rx); micromoles per liter (µmol/L); millimoles per liter (mmol/L); grams per liter (g/L); Units per liter (U/L); Aspartate Aminotransferase (AST); Blood Urea Nitrogen (BUN) Total Bilirubin: >1.1*ULN if Pre-Rx<= ULN or Pre-Rx is missing, or >1.2*Pre-Rx if Pre-Rx >ULN. AST: >1.25*Pre-Rx if Pre-Rx >ULN or 1.25*ULN if Pre-Rx <= ULN or Pre-Rx is missing. BUN: >1.1*ULN if Pre-Rx<= ULN or Pre-Rx is missing, or >1.2*Pre-Rx if Pre-Rx >ULN. Phosphorus: <0.85*LLN if Pre-RX >= LLN or is missing or if Pre-Rx < LLN. total Protein: <0.9*LLN if Pre-Rx>= LLN or is missing or Pre-Rx > LLN. Creatine Kinase: >1.5*Pre-Rx if Pre-Rx > ULN or is missing or Pre-Rx is <= ULN. Lactate Dehydrogenase: >1.25*ULN if Pre-Rx <= ULN or missing, >1.5*Pre-Rx if Pre-Rx > ULN.
Time Frame: Day -1 to Day 46 ±2 days or at early termination
Population: Participants who received any study medication and had laboratory test results.
Measure: Number; unit: participants
Arm/Group | Inje Cocktail Alone and Inje Cocktail Plus Belatacept
Number analyzed (Participants) | 22
participants
  Total bilirubin >1.1*ULN µmol/L (N=22) | 1
  AST >1.25*Pre-Rx U/L (N=22) | 1
  BUN >1.1*ULN mmol/L (N=22) | 1
  Inorganic Phosphorus <0.85*LLN mmol/L (N=22) | 1
  Total Protein <0.9*LLN g/L (N=22) | 1
  Creatine Kinase > 1.5* Pre-Rx U/L (N=22) | 2
  Lactate Dehydrogenase >1.25*ULN U/L (N=22) | 1

31. Secondary Outcome: Number of Participants With Marked Hematology and Urinalysis Laboratory Abnormalities - All Treated Participants
Description: Samples for laboratory tests were obtained at Screening visit, Day -1 or prior to dosing on Day 1, Days 3, 6, 10, 46 ±2, and at early termination, after 10 hours fasting. Leukocytes: *10^9 cells per liter (c/L) < 0.85*Pre-Rx if Pre-Rx < LLN or <0.9*LLN if LLN <= Pre-Rx or Pre-Rx is missing. Neutrophils (absolute): *10^12 c/L < 0.85* Pre-Rx if Pre-Rx < 1.5, <1.5 if Pre-Rx >= 1.5, < 1.5 if Pre-Rx missing. Urine blood from dipstick: >=2 if Pre-Rx <1 or was missing or if Pre-Rx >=1. Urinary microscopic white blood cells (WBC) and red blood cells (RBC) >= 2 if Pre-Rx <2 or if Pre-Rx was missing or >=4 if Pre-Rx >=2.
Time Frame: Day -1 to Day 46 ±2 days or at early termination
Population: Participants who received any study medication and had laboratory test results.
Measure: Number; unit: participants
Arm/Group | Inje Cocktail Alone and Inje Cocktail Plus Belatacept
Number analyzed (Participants) | 22
participants
  Leukocytes <0.85*Pre-Rx *10^9 c/L (N=22) | 1
  Neutrophils <0.85*Pre-Rx *10^12 c/L (N=22) | 4
  Urine Blood >= 2 (N=22) | 2
  Urinary RBC microscopic >= 2 (N=8) | 1
  Urinary WBC microscopic >= 2 (N=8) | 1

32. Secondary Outcome: Number of Participants With Out-of-Range Electrocardiogram Intervals - All Treated Participants
Description: Participants had 12-Lead electrocardiograms (ECGs) performed at Screening Visit, Day 1 prior to dosing, Day 46 ±2, and at early termination. Definition of out-of-range: PR Interval >210 milliseconds (msec); QRS > 120 msec, QT > 500 msec or > 30 msec change from baseline (Day 1); QT with Fridericia correction (QTcF) > 450 msec or change from baseline of > 30 msec to <= 60 msec or change from baseline > 60 msec.
Time Frame: Day 1 to Day 46 ±2 days or at early termination
Population: All participants who received any study medication and had an ECG performed on Day 1, Day 46 or early termination.
Measure: Number; unit: participants
Arm/Group | Inje Cocktail Alone and Inje Cocktail Plus Belatacept
Number analyzed (Participants) | 18
participants
  Day 46 (N=18) | 0
  Early Termination (N=2) | 0

33. Secondary Outcome: Mean Change From Baseline in Sitting Systolic and Diastolic Blood Pressure - All Treated Participants
Description: Systolic and Diastolic blood pressures were taken after the participant had been sitting quietly for at least 5 minutes and the pressures were measured in millimeters of mercury (mm Hg). Pressures were obtained at screening visit, Day -1, and at 0 hour (pre-dose), 0.5 hour (post dose), and 2 hours (post dose) on Days 1, 4, 7, 11. Baseline was defined as last non-missing result with a collection date-time less than the date-time of the first active dose of study drug.
Time Frame: Baseline and 0.5 and 2.0 hours Post Dose on Days 1, 4, 7, and 11
Population: All participants who received any study medication and had a baseline and specific day blood pressure measurement available.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
mm Hg
  Systolic 0.5 hour post dose (N=22,21,21,20) | -0.6 (10.15) | 0.1 (12.81) | -4.9 (9.05) | -4.7 (10.13)
  Systolic 2.0 hour post dose (N=22,21,21,20) | 0.2 (10.09) | 2.0 (11.79) | -2.7 (9.85) | -2.9 (11.73)
  Diastolic 0.5 hour post dose (N=22,21,21,20) | -1.7 (6.52) | -0.2 (6.03) | -2.2 (7.54) | -2.2 (5.38)
  Diastolic 2.0 hour post dose (N=22,21,21,20) | 0.9 (4.67) | -2.0 (4.53) | -3.4 (5.22) | -1.0 (5.83)

34. Secondary Outcome: Mean Change From Baseline in Sitting Heart Rate - All Treated Participants
Description: Heart Rate was taken after the participant had been sitting quietly for at least 5 minutes and the heart rate was measured in beats per minute (bpm). Heart Rates were obtained at screening visit, Day -1, and at 0 hour (pre-dose), 0.5 hour (post dose), and 2 hours (post dose) on Days 1, 4, 7, 11. Baseline was defined as last non-missing result with a collection date-time less than the date-time of the first active dose of study drug.
Time Frame: Baseline and 0.5 and 2.0 hours Post Dose on Days 1, 4, 7, and 11
Population: All participants who received study medication and had baseline and specific day measurement.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Day 1 Inje Cocktail | Day 4 Inje Cocktail Plus Belatacept | Day 7 Inje Cocktail | Day 11 Inje Cocktail
Number analyzed (Participants) | 22 | 21 | 21 | 20
bpm
  Heart Rate 0.5 hour post dose (N=22, 21, 21, 20) | -3.3 (12.38) | -4.2 (13.15) | -1.8 (12.58) | -1.6 (10.03)
  Heart Rate 2.0 hour post dose (N=22, 21, 21, 20) | -3.5 (10.61) | 0.2 (13.86) | 0.5 (11.95) | 3.1 (11.91)

35. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure at Study Discharge (Day 46±2 Days)
Description: Systolic and Diastolic blood pressures were taken after the participant had been sitting quietly for at least 5 minutes and the pressures were measured in millimeters of mercury (mm Hg). Systolic and Diastolic blood pressures were taken on Day 46 (day of discharge from the study). Baseline was defined as last non-missing result with a collection date-time less than the date-time of the first active dose of study drug.
Time Frame: Baseline and Day 46 ±2 days
Population: All participants who had received study drug during the treatment period and had measurements at baseline and at discharge.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Post Treatment: Days 12 through 46 (Day of Discharge from Study). No study drug was administered during this time.
Arm/Group | Post Treatment
Number analyzed (Participants) | 18
mm Hg
  Systolic (N=18) | -5.9 (11.25)
  Diastolic (N=18) | -5.7 (8.87)

36. Secondary Outcome: Mean Change From Baseline in Heart Rate at Study Discharge (Day 46±2 Days)
Description: Heart Rate was taken after the participant had been sitting quietly for at least 5 minutes and was measured in beats per minute (bpm). Hear rate was taken on Day 46 (day of discharge) during the follow up period. Baseline was defined as last non-missing result with a collection date-time less than the date-time of the first active dose of study drug.
Time Frame: Baseline and Day 46 ±2 days
Population: All participants who received study drug during the treatment period and had measurements at baseline and discharge.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Post Treatment
Number analyzed (Participants) | 18
bpm | 1.0 (15.86)

ADVERSE EVENTS:
Time Frame: Day 1 to Day of discharge (Day 46 ±2 days)
Arm/Group | Inje Cocktail Alone and Inje Cocktail Plus Belatacept
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inje Cocktail Alone and Inje Cocktail Plus Belatacept (N=22)
Headache (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.